CLINICAL TRIAL: NCT03952767
Title: The STEPP Study: Sensors To Evaluate Physical Performance
Acronym: STEPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LCCC 1851
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Physical Measures and Survey Assessments (Experimental): Digital physical measure data will be collected in clinic and at home and survey assessments will be collected
  Interventions: Other: Digital Physical Measures and Survey Assessments

INTERVENTIONS:
Other: Digital Physical Measures and Survey Assessments — Data from at home and in clinic visits will assess physical function and survey data will be collected

SUMMARY:
This study assesses the association between digital functional measures of physical and patient-reported standard onocological assessments, like Karnofsky Performance Score (KPS).

DETAILED DESCRIPTION:
This study assess the association between digital functional measures from physical monitoring devices (devices like a watch tracking steps, a heart rate monitor) and patient-reported standard oncological assessments. The study will also test the feasibility of obtaining the measures in clinic and at home from the monitoring devices in participants with cancer. Participants will be asked to spend 1 hour in clinic performing simple tasks such as walking and standing with 7 digital devices recording movement data. The participants will also be asked to fill out survey data regarding their health. At-home data will be collected for 14 days. During this time participants will wear a watch to collect movement and step data, and a lumbar belt to collect movement data.

Primary Objective:

1. Assess the association of 5 main digital physical functional measures (mean steps per day, mean sedentary activity time, light activity time, moderate activity time, and vigorous activity time (in minutes) per day) recorded at home with patient-reported standard oncological assessment (e.g. KPS)

ELIGIBILITY:
Inclusion Criteria:

1. All genders aged ≥ 18 years of age
2. Patients being seen at UNCCH for treatment of cancer.
3. English-speakers
4. Able to understand and cooperate with study procedures.
5. Patients with solid tumors or hematological malignancies, and self-reported KPS ≤70 to ≥ 100.

Signed and dated informed consent and HIPPA.

Exclusion Criteria:

1. Subjects using investigational/experimental products.
2. Has dementia, altered mental status, or any psychiatric or co-morbid condition prohibiting the understanding or rending of informed consent.
3. Unable or unwilling to complete physical performance assessments including the at-home wearable device for 14 days.
4. Unable to speak English.
5. Subjects who report any other medical condition, recreational substance use, or medication use which would prevent them from completing study tasks or impair the providing of informed consent.
6. Subjects who are allergic to silicone or adhesives. Subjects with cardiac pacemakers, electronic pumps or any other implanted medical devices.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Amount of mean steps per day recorded at home | 18 months
  At-home record of mean steps per day
Amount of mean sedentary activity time recorded at home | 18 months
  At-home record of minutes per day of mean sedentary activity time
Amount of Light activity time recorded at home | 18 months
  At-home record of minutes per day of light activity time per day
Amount of moderate activity time recorded at home | 18 months
  At-home record of minutes per day of moderate activity time
Amount of vigorous activity time recorded at home | 18 months
  At-home record of minutes per day of vigorous activity time
Self-Reported Karnofsky Performance Score (KPS) | 18 months
  The validated 1 question Self-reported Karnofsky Performance Score (KPS) score 0 to 100 will be measured. Scores closer to 100 indicate high performance of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karahanoglu FI, Jensen CE, Cai X, Santamaria M, Psaltos D, Messere A, Demanuele C, Stone J, Tarachandani A, Adamowicz L, Muss H, Wood WA. Improved functional assessment in cancer patients using home-based digital technologies. Sci Rep. 2025 May 21;15(1):17638. doi: 10.1038/s41598-025-02401-4. PMID 40399391